CLINICAL TRIAL: NCT05465694
Title: The Role of Time Interval Elimination on Pain Control of Preterm Infants by Sucrose Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Deniz Yaprak, Director, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEAH.Denizyaprak.137470
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Neonatal Disease; Pain, Acute
Keywords: preterm; pain; sucrose; dopamine
MeSH Terms: conditions — Infant, Newborn, Diseases; Acute Pain; Premature Birth; Pain | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-minute-time interval of per oral 24% sucrose (Active Comparator): For infants in the 2-minute-time interval of per oral 24% sucrose was given prior to the heel lance intervention.
  Interventions: Procedure: 2-minute-time interval of per oral 24% sucrose
- no time interval of per oral 24% sucrose (Active Comparator): In no time interval of sucrose was given immediately prior to heel lance intervention.
  Interventions: Procedure: no time interval of per oral 24% sucrose

INTERVENTIONS:
Procedure: 2-minute-time interval of per oral 24% sucrose — Experiment began with a five-minute observation period of all outcome measures while infant was resting in an incubator. Later, attendant nurse gave 1 ml of 24% sucrose solution on neonate's tongue. In the 2-two minute-time interval prior to heel lance intervention, following two minutes of waiting period, heel lance procedure was applied to infant's foot. In no time interval of sucrose given immediately prior to heel lance intervention, attendant nurse performed heel lance procedure immediately after giving 1 ml of 24% sucrose solution sucrose on tongue. Infant's facial actions and heart rate, and oxygen saturation were recorded by using two video cameras. Recording was carried out by a nurse during whole procedure. After collecting data, researcher watched videos separately and scored them by using PIPP-R. Measurement of study outcome relied on data collection strategies: Neonatal close-up video recording of infant facial actions, pulse oximeter, observation for adverse events.
  Arms: 2-minute-time interval of per oral 24% sucrose
Procedure: no time interval of per oral 24% sucrose — no time interval of per oral 24% sucrose
  Arms: no time interval of per oral 24% sucrose

SUMMARY:
Purpose. It has been demonstrated clearly that sucrose solutions given before a minor painful procedure can reduce pain among newborns. But, there are no entirely accepted conclusions about the time scheduling of sucrose administration prior to heel lance. In a few studies, various time intervals between sucrose intake and heel lance procedure have been proposed. The aim of this study was to obtain a deeper knowledge of the underlying mechanism by investigating whether a different initiation of heel lance in terms of timing would reduce the effect of orally administered sucrose at heel lance among preterm newborns.

Methods. A randomized, double-blind trial with a validated, neonatal, pain-scoring scale in Gulhane Medical School Hospital in Ankara, Turkey between March 2019 and January 2021. The trial included 69 preterm newborns undergoing heel lance, who were assigned randomly to 1 of 2 groups, ie, group I, with the 2-minute-time interval of per oral 24% sucrose given prior to heel lance or group II, without a time interval of per oral sucrose given prior to heel lance. Pain-related behavior during blood sampling was measured with the Premature Infants Pain Profile-Revised (PIPP-R). Crying incidence, duration, and heart rate were also recorded. The aim of this study was to help to clarify the mechanism underlying the pain-reducing effect of orally administered sucrose by attempting to determine whether elimination of the time interval prior to heel lance would reduce the effect of oral sucrose among preterm newborns. Investigators hypothesized that there would be a significant difference in pain intensity without a waiting period after sucrose ingestion, measured at 30 and 60 s following heel lance using PIPP-R, and adverse events would be higher.

DETAILED DESCRIPTION:
The sample size was calculated based on the difference in the PIPP scores of the groups. A sample size of 54 (27 for each group) achieves 80% power to detect a large effect size of 0.8 using a two-sided Mann-Whitney U test with a significance level of 0.05.

After inclusion in the study, participating infants were randomized to one of two possible interventions during a clinically-required heel lance: 1) The 2-minute-time interval of per oral 24% sucrose given prior to heel lance (Group 1) or no time interval of per oral 24% sucrose given prior to heel lance (Group 2) combined with containment in a blanket while in an infant incubator. Enrollment and randomization into the 2-minute-time interval of per oral 24% sucrose given prior to heel lance or no time interval of per oral 24% sucrose given prior to heel lance (within 10 s) interventions were carried out by a member of the research team using a computerized off-site password protected website. Intervention allocation concealment was achieved by using randomly permuted stratified randomization of gestational week and gender. The treatment allocations were inserted into identical sealed envelopes marked only with a number. Solutions of 24% sucrose were freshly prepared daily by pharmacy using 2.4 g sucrose plus 10 ml distilled water. Solutions were packaged in 1 ml sterile syringes and further packaged in opaque sealed envelopes labeled according to the randomization code. The research team including two clinicians and nurses were masked in the treatment allocation. Outcome assessor was also blinded.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are premature born ( ≥ 27 0/7 weeks of gestation)
* Infants who are at the postconceptional age from 34 0/7- 37 6/7 weeks of gestation
* Normal enterally fed with human milk or formula
* Infants whose mothers consented to study participation

Exclusion Criteria:

* Infants who were born depressed or with birth trauma
* Infants who have previous surgery
* Infants who have an intraventricular hemorrhage
* Infants who show signs of respiratory distress
* Infants who have an infection
* Infants with significant genetic disorders
* Infants who were on sedatives, muscle relaxants, and antiepileptic
* Infants who were born to opioid-using mothers
* Infants whose parents were unable to provide written informed consent

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile-Revised (PIPP-R) | 30 seconds
  The PIPP-R is a seven indicator composite pain measure consisting of three behavioural (facials actions of brow bulge, eye squeeze, naso-labial furrow), two physiological (heart rate, oxygen saturation), and two contextual (gestational age, behavioural state) indicators validated for pain measurement in infants 26-44 weeks' gestation. A score of <7 is indicative of minimal pain and a score ≥ 12 is indicative of moderate to severe pain.
Premature Infant Pain Profile-Revised (PIPP-R) | 60 seconds
  The PIPP-R is a seven indicator composite pain measure consisting of three behavioural (facials actions of brow bulge, eye squeeze, naso-labial furrow), two physiological (heart rate, oxygen saturation), and two contextual (gestational age, behavioural state) indicators validated for pain measurement in infants 26-44 weeks' gestation. A score of <7 is indicative of minimal pain and a score ≥ 12 is indicative of moderate to severe pain.

SECONDARY OUTCOMES:
Crying incidence | 120 seconds
  The proportion of infants who cry during the heel lance procedure
Crying duration | 120 seconds
  The mean crying time in infants who cry
Heart rate | 30 seconds
  The mean heart beat rate in a minute
Heart rate | 60 seconds
  The mean heart beat rate in a minute

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Yaprak, MD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Gulhane Medicine Faculty, Department of Pediatrics, Division of Neonatology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After acceptance of the trial registry, the director is going to decide to make individual participant data (IPD) available to other researchers.